CLINICAL TRIAL: NCT02553733
Title: Effects of Dietary Nitrate Supplementation on Coronary Blood Flow and Walking Performance in Peripheral Arterial Disease
Brief Title: Effect of Beetroot Juice on Coronary Blood Flow and Walking Performance in PAD
Acronym: HeartBeet
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: David N. Proctor, PhD (Other)
Collaborators: Milton S. Hershey Medical Center (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor-Investigator, David N. Proctor, PhD, Professor of Kinesiology and Physiology, Penn State University
Organization: Penn State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 00003242
Record Dates: First submitted 2015-09-15; First posted 2015-09-18 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Peripheral Arterial Disease
Keywords: Dietary nitrate supplementation; Beetroot juice
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Beetroot juice (Beet-It Organic Shot) (Active Comparator): Subjects will consume 70 ml of beetroot juice (Beet-It Organic Shot) twice per day (morning, afternoon) for 5 to 7 days to assess the short term effects of this nitrate supplement on graded treadmill walking responses (day 4) and vasodilator/vasoconstrictor responses in the coronary and lower leg circulations (day 5 or 6 or 7). On both study visits, subjects will consume their morning dose 1 hour 45 min before experiments begin.
  Interventions: Drug: Beetroot juice
- Beetroot juice placebo (Beet-It Organic Placebo) (Placebo Comparator): Subjects will consume 70 ml of beetroot juice placebo (Beet-It Organic Placebo) twice per day (morning, afternoon) for 5 to 7 days to assess the short term effects of this nitrate supplement on graded treadmill walking responses (day 4) and vasodilator/vasoconstrictor responses in the coronary and lower leg circulations (day 5 or 6 or 7). On both study visits, subjects will consume their morning dose 1 hour 45 min before experiments begin.
  Interventions: Drug: Beetroot juice placebo

INTERVENTIONS:
Drug: Beetroot juice — This beverage contains 0.3 g of inorganic nitrate per 70 ml container, and is bottled and supplied by James White Drinks (UK).
  Other Names: Beet-It Organic Shot
  Arms: Beetroot juice (Beet-It Organic Shot)
Drug: Beetroot juice placebo — This beverage is identical in look and taste to the Beet-It organic shot, but has the nitrate removed. It is also bottled and supplied by James White Drinks (UK).
  Other Names: Beet-It organic placebo
  Arms: Beetroot juice placebo (Beet-It Organic Placebo)

SUMMARY:
In this study the investigators will test the hypothesis that short-term consumption of inorganic nitrate (supplied in concentrated beetroot juice) enhances coronary blood flow responses, large artery hemodynamics, and leg oxygenation/exercise tolerance in patients with peripheral arterial disease (PAD). Understanding and improving blood flow regulation in the heart and skeletal muscles of patients with PAD is important because exercise triggers symptoms of leg pain and substantially raises blood pressure and myocardial demand in these patients.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is a strong predictor of cardiovascular mortality and negatively affects functional capacity and quality of life for as many as 14 million patients in the U.S. alone. One open-label study showed that acute consumption of beetroot juice improved 6 min walk performance, reduced blood pressure, and enhanced leg muscle oxygenation in PAD patients. However, no studies have rigorously confirmed these findings in a double-blind manner, nor have the effects of this supplement been investigated (acutely or short-term) in the coronary circulation of PAD patients.

In addition to studying its effects on graded treadmill walking performance and consequent large artery vasodilation, the present study will examine the effects of short-term beetroot juice consumption (twice/day) on both coronary and leg vasodilator (graded calf flexion) and vasoconstrictor (isometric handgrip, voluntary apnea) responses in patients with PAD. Participants will randomly consume either nitrate-rich or nitrate-depleted beetroot juice with a 7 to 14 day wash-out period between. Effects of beetroot juice consumption on plasma nitrate, nitrite and methemoglobin will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with peripheral arterial disease (PAD)
2. Capable of giving informed consent
3. Men and women age 21- 85 years
4. Diagnosed with PAD (i.e., ankle-brachial index below 0.9)
5. Fontaine stage II or less - no pain while resting
6. Satisfactory history and physical exam

Exclusion Criteria:

1. Children
2. Pregnant or nursing women
3. Patients taking nitroglycerine or nitrate preparations
4. Patients taking phosphodiesterase inhibitors such as sildenafil or tadalafil
5. Patients taking proton pump inhibitors
6. Ejection fraction < 40%
7. Uncontrolled hypertension
8. Uncontrolled diabetes
9. Myocardial infarction within past 6 months or unstable angina
10. Severe lung disease (i.e., on supplemental oxygen or frequently use rescue inhalers)
11. Abnormality in hemoglobin or hematocrit or methemoglobin
12. Impaired renal function
13. Impaired liver function
14. History or diagnosis of Barrett's esophagus
15. Known allergy to beetroot juice or lemon juice
16. Inability to walk on a treadmill at a moderate pace (2.0 miles/hour)

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-12; Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Exercise performance | 5 to 7 days after initiating daily ingestion of beetroot juice
  Exercise capacity will be assessed using a graded treadmill walking test to peak exertion with expired gas analysis and determination of peak oxygen uptake, calf muscle oxygenation, blood pressure, claudication onset time, and peak walking time.

SECONDARY OUTCOMES:
Coronary vascular function | 4 days after initiating daily ingestion of beetroot juice
  Coronary artery (transthoracic ultrasound) blood flow responses to plantar flexion and handgrip exercise.
Leg vascular function | 4 days after initiating daily ingestion of beetroot juice
  Popliteal artery and near infrared spectroscopy (NIRS) responses to plantar flexion and handgrip exercise.

OTHER OUTCOMES:
Blood measures of nitrate absorption and conversion | 4 to 7 days after initiating ingestion of beetroot juice
  Venous blood will be withdrawn (venipuncture) for determination of plasma nitrate, nitrite and methemoglobin levels

CONTACTS AND LOCATIONS:
Overall Officials: Urs A Leuenberger, MD, Principal Investigator — Penn State University
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Kim DJ, Gao Z, Luck JC, Brandt K, Miller AJ, Kim-Shapiro D, Basu S, Leuenberger U, Gardner AW, Muller MD, Proctor DN. Effects of short-term dietary nitrate supplementation on exercise and coronary blood flow responses in patients with peripheral artery disease. Front Nutr. 2024 Jul 3;11:1398108. doi: 10.3389/fnut.2024.1398108. eCollection 2024. PMID 39027664